CLINICAL TRIAL: NCT01664728
Title: An Expanded Access Open Label Study of CB7630 (Abiraterone Acetate) in Patients With Advanced Prostate Cancer Who Have Completed CB7630 Clinical Study COU-AA-001
Brief Title: An Expanded Access Study of Abiraterone Acetate in Patients With Advanced Prostate Cancer Who Have Completed Clinical Study COU-AA-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016912; COU-AA-001EXT (Other: Janssen Research & Development, LLC); 2006-006755-12 (EudraCT Number)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Hormone refractory prostate cancer; Castration resistant prostate cancer; Castration refractory prostate cancer; Abiraterone acetate; CB7630
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate (Experimental)
  Interventions: Drug: Abiraterone acetate; Drug: Glucocorticoid

INTERVENTIONS:
Drug: Abiraterone acetate — Phase 2 maximum tolerated dose from Study COU-AA-001 taken orally once daily
Drug: Glucocorticoid — prednisolone/prednisone 5 mg taken orally twice daily or dexamethasone 0.5 mg taken orally once daily

SUMMARY:
The purpose of this study is to provide access to abiraterone acetate for patients who have completed 12 cycles of abiraterone acetate treatment in Clinical Study COU-AA-001 and continue to receive clinical benefit from this treatment.

DETAILED DESCRIPTION:
This is an open-label (identity of study drug will be known) extended access study to evaluate the safety and efficacy of continued administration of abiraterone acetate in patients who have completed 12 cycles of abiraterone acetate treatment in Clinical Study COU-AA-001 and continue to receive clinical benefit from this treatment. Patients will continue with the same dose regimen administered at the end of Study COU-AA-001 and will receive a low-dose glucocorticoid daily. Patients will be followed every 3 months for disease progression and survival for up to 3 years following study entry. Safety will be monitored throughout the study up to 30 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Completed 12 cycles of abiraterone acetate under study COU-AA-001
* Last dose of abiraterone acetate within 14 days prior to treatment in this study
* Demonstrates potential to gain clinical benefit with continued abiraterone acetate treatment
* Serum potassium level >=3.5 mmol/L
* Eastern Cooperative Oncology Group Performance Status of <3 (Karnofsky Performance Status >=30%)
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Uncontrolled hypertension
* Abnormal liver function
* Clinically significant heart disease as evidenced by a myocardial infarction in the past 12 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease (patients with a history of atherosclerotic vascular disease requiring coronary or peripheral artery bypass surgery may be enrolled provided the surgery occurred at least 2 years prior to enrollment and after consultation with a cardiologist to insure that the disease is stable)
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with serum prostate specific antigen (PSA) decline according to PSA Working Group criteria | Screening, Cycle 1 Day 1 Pre-dose, every 3 months up to 3 years after study entry
Overall survival | every 3 months up to 3 years after study entry

SECONDARY OUTCOMES:
Number of participants with adverse events | up to 30 days after the last dose of study medication
Time to disease progression | every 3 months up to 3 years after study entry
Time to prostate specific antigen progression | every 3 months up to 3 years after study entry
Objective tumor response by Response Evaluation Criteria in Solid Tumors (RECIST) | every 3 months up to 3 years after study entry

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Sutton, United Kingdom

REFERENCES:
- See also: An Expanded Access Open Label Study of CB7630 (Abiraterone Acetate) in Patients with Advanced Prostate Cancer Who Have Completed CB7630 Clinical Study COU-AA-001 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2388&filename=CR016912_CSR.pdf